CLINICAL TRIAL: NCT01536522
Title: Asthma Inflammation Research
Acronym: AIR
Status: Enrolling by invitation | Phase: Early Phase 1 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Serpil Erzurum, Chair of Lerner Research Institute, The Cleveland Clinic
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Other
Other Study IDs: 10-1049; PAR-09-185 (Other: NIH)
Record Dates: First submitted 2012-02-13; First posted 2012-02-22 (Estimated); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Asthma; Allergic Asthma; Non-allergic Asthma
Keywords: Asthma; Allergic Asthma; Non-allergic Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: feasibility and palatability of a food product for asthma
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Nutritional Approach for Asthma (Active Comparator): individuals will be provide a pre measured dose of medium chain triglyceride to consume along with their meals. They will be instructed to add the MCT to their meal 3 times per day
  Interventions: Dietary Supplement: Nutritional approach for asthma
- Standard American Diet (Placebo Comparator): patients will consume their usual diet with a pre measured dose of canola oil in place of the medium chain triglyceride as a control group. They will be instructed to add the placebo dose to their meal 3 times a day
  Interventions: Dietary Supplement: Nutritional approach for asthma
- Alternate Day Diet (Active Comparator): patients will consume a regular "Standard American Diet" for 4 weeks and then provided a regulated dosed quantity of low caloric value "shakes". they will consume this on alternating days
  Interventions: Dietary Supplement: Low Caloric Shake
- Whole Lung Allergen Challenge (Active Comparator): patients with or without asthma will be given controlled doses of specified allergens
  Interventions: Biological: whole lung allergen challenge

INTERVENTIONS:
Dietary Supplement: Nutritional approach for asthma — participants will be provided a medium chain triglyceride supplement or placebo
  Other Names: MCT supplement
  Arms: Nutritional Approach for Asthma; Standard American Diet
Dietary Supplement: Low Caloric Shake — participants will be provided a low caloric dietary shake
  Arms: Alternate Day Diet
Biological: whole lung allergen challenge — inhalation of allergens by allergic patients with or without asthma, will be used to define mechanisms underlying the development of airway inflammation
  Arms: Whole Lung Allergen Challenge

SUMMARY:
The overall goal of the Asthma Inflammation Research [AIR] Translational Program is to create an integrated multidisciplinary team for the focused purpose of development of diagnostic and prognostic tests informative for airway inflammation, and for the design of innovative, targeted biologic therapeutics.

The overarching aims of the AIR program are to conceptualize, develop, and test the next-generation therapeutics, and novel asthma diagnostic and prognostic tools that will allow us to improve the standard of asthma care.

DETAILED DESCRIPTION:
More than 20 million Americans suffer from asthma, and nearly half of asthma sufferers do not have their asthma under control. Although commonly diagnosed using physiological measures of airflow and bronchial hyperreactivity, asthma pathophysiology is related to chronic inflammation of the airway.

Current diagnostic evaluation and monitoring are inadequate for proposed practice guidelines. The most commonly used test for evaluation of asthma is the measurement of airflow obstruction by spirometry. The National Asthma Education Prevention Program (NAEPP) and Expert Panel Reports set forth grading of asthma severity based on the frequency of symptoms, airflow, and the need for inhaled beta-agonists. Practice guidelines outline that the goals of therapy for asthma are to: maintain normal activity with near normal parameters of lung function, prevent exacerbations that lead to tissue injury, and avoid medication toxicity. In order to facilitate these goals, NAEPP defines key components for management including disease monitoring and stepped care pharmacotherapy. Unfortunately, there is no optimal plan for monitoring inflammation, which causes us to fail in key components in management of asthma. Limited options for anti-inflammatory treatments to control asthma likewise often lead to substantial morbidities due to treatment with high doses of corticosteroids. Our AIR program plans to develop novel asthma monitoring tests and design targeted therapeutics, which altogether may reduce toxicities and improve the long-term health of patients.

Impact on broad scientific advancement. Our cumulative studies provide fundamental information on the molecular mechanisms that contribute to unresolving and excessive inflammation that leads to tissue remodeling. This mechanistic knowledge is of broad scientific importance as nearly all chronic human diseases are defined by prolonged and active inflammation, with tissue destruction, and failed attempts at healing. Thus, our investigations will provide comprehensive knowledge and consequent translational deliverables that may be widely applicable as diagnostic strategies and therapies in other chronic inflammatory diseases.

ELIGIBILITY:
Inclusion Criteria:

* Asthma diagnosed by a medical specialist and/or history of positive methacholine rest and/or reversibility of >10% of FEV1
* FEV1 is within acceptable limits
* Informed Consent is present

Exclusion Criteria:

* Diabetes (fasting blood sugar >110 mg/dL)
* Any milk allergies
* Coconut allergies
* BMI >40 kg/m2,
* Inability to maintain diet intervention
* Current smoking or smoking history of greater than 10 pack-years
* Any other significant respiratory or cardiac disease or the presence of clinically important comorbidities, including, uncontrolled coronary artery disease, acute or and chronic renal failure

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Maintaining a tolerance to Medium Chain Triglyceride (MCT) additive for Asthmatics | 24 weeks
  Tolerability of the MCT will be assessed by maintenance of use of MCT by 20% or more participants over the 3 months of the study.

SECONDARY OUTCOMES:
Improvement of lung function by spirometry testing | 24 weeks
  Quantitative data will be collected to evaluate any improvement mechanistically in the lungs using breathing tests
Asthma Quality of Life Questionnaire | 24 weeks
  Asthma Quality of Life Questionnaire will be evaluated for any decrease in asthma symptoms by a 7 point scale. 7 is not impaired and 1 is severely impaired. The higher the total score will determine better quality of life
Asthma Control Test | 24 weeks
  Asthma control test will be used to score improvement in day to day activities using a 5 point lscale. A score of 1 equals all of the time and a score of 5 equals not at all. The score ranges of 5 (poorly controlled) to 25 (complete control). A total ACT score greater than 19 indicates asthma is well controlled
Gastrointestinal tolerance of a Medium Chain Triglyceride additive to a normal diet in Asthmatics | 12
  GI symptoms will be documented and data captured to measure tolerance via a 5 point scale. A score of 1 equals symptoms all of the time and 5 equals never. The greater the score indicates less or no GI symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Serpil Erzurum, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

REFERENCES:
- [Background] National Asthma Education and Prevention Program. National Asthma Education and Prevention Program. Expert Panel Report: Guidelines for the Diagnosis and Management of Asthma Update on Selected Topics--2002. J Allergy Clin Immunol. 2002 Nov;110(5 Suppl):S141-219. No abstract available. PMID 12542074
- [Background] National Asthma Education and Prevention Program. Expert Panel Report 3 (EPR-3): Guidelines for the Diagnosis and Management of Asthma-Summary Report 2007. J Allergy Clin Immunol. 2007 Nov;120(5 Suppl):S94-138. doi: 10.1016/j.jaci.2007.09.043. PMID 17983880
- [Background] Dweik RA, Sorkness RL, Wenzel S, Hammel J, Curran-Everett D, Comhair SA, Bleecker E, Busse W, Calhoun WJ, Castro M, Chung KF, Israel E, Jarjour N, Moore W, Peters S, Teague G, Gaston B, Erzurum SC; National Heart, Lung, and Blood Institute Severe Asthma Research Program. Use of exhaled nitric oxide measurement to identify a reactive, at-risk phenotype among patients with asthma. Am J Respir Crit Care Med. 2010 May 15;181(10):1033-41. doi: 10.1164/rccm.200905-0695OC. Epub 2010 Feb 4. PMID 20133930
- [Background] Crapo RO, Morris AH, Gardner RM. Reference spirometric values using techniques and equipment that meet ATS recommendations. Am Rev Respir Dis. 1981 Jun;123(6):659-64. doi: 10.1164/arrd.1981.123.6.659. PMID 7271065
- [Background] Standardization of Spirometry, 1994 Update. American Thoracic Society. Am J Respir Crit Care Med. 1995 Sep;152(3):1107-36. doi: 10.1164/ajrccm.152.3.7663792. No abstract available.
- [Background] Hankinson JL, Odencrantz JR, Fedan KB. Spirometric reference values from a sample of the general U.S. population. Am J Respir Crit Care Med. 1999 Jan;159(1):179-87. doi: 10.1164/ajrccm.159.1.9712108. PMID 9872837
- [Background] Juniper EF, Guyatt GH, Epstein RS, Ferrie PJ, Jaeschke R, Hiller TK. Evaluation of impairment of health related quality of life in asthma: development of a questionnaire for use in clinical trials. Thorax. 1992 Feb;47(2):76-83. doi: 10.1136/thx.47.2.76. PMID 1549827
- [Background] Dweik RA, Comhair SA, Gaston B, Thunnissen FB, Farver C, Thomassen MJ, Kavuru M, Hammel J, Abu-Soud HM, Erzurum SC. NO chemical events in the human airway during the immediate and late antigen-induced asthmatic response. Proc Natl Acad Sci U S A. 2001 Feb 27;98(5):2622-7. doi: 10.1073/pnas.051629498. Epub 2001 Feb 20. PMID 11226289
- [Background] Dweik RA, Lewis M, Kavuru M, Buhrow L, Erzurum SC, Thomassen MJ. Inhaled corticosteroids and beta-agonists inhibit oxidant production by bronchoalveolar lavage cells from normal volunteers in vivo. Immunopharmacology. 1997 Oct;37(2-3):163-6. doi: 10.1016/s0162-3109(97)00043-x. PMID 9403334
- [Background] Dweik RA, Mehta AC, Meeker DP, Arroliga AC. Analysis of the safety of bronchoscopy after recent acute myocardial infarction. Chest. 1996 Sep;110(3):825-8. doi: 10.1378/chest.110.3.825. PMID 8797432
- [Background] Dweik RA, Stoller JK. Role of bronchoscopy in massive hemoptysis. Clin Chest Med. 1999 Mar;20(1):89-105. doi: 10.1016/s0272-5231(05)70129-5. PMID 10205720
- [Background] American Thoracic Society; European Respiratory Society. ATS/ERS recommendations for standardized procedures for the online and offline measurement of exhaled lower respiratory nitric oxide and nasal nitric oxide, 2005. Am J Respir Crit Care Med. 2005 Apr 15;171(8):912-30. doi: 10.1164/rccm.200406-710ST. No abstract available. PMID 15817806
- [Background] Khatri SB, Hammel J, Kavuru MS, Erzurum SC, Dweik RA. Temporal association of nitric oxide levels and airflow in asthma after whole lung allergen challenge. J Appl Physiol (1985). 2003 Jul;95(1):436-40; discussion 435. doi: 10.1152/japplphysiol.01127.2002. Epub 2003 Feb 7. PMID 12576414
- [Background] Khatri SB, Ozkan M, McCarthy K, Laskowski D, Hammel J, Dweik RA, Erzurum SC. Alterations in exhaled gas profile during allergen-induced asthmatic response. Am J Respir Crit Care Med. 2001 Nov 15;164(10 Pt 1):1844-8. doi: 10.1164/ajrccm.164.10.2106119. PMID 11734434
- [Background] Wu W, Samoszuk MK, Comhair SA, Thomassen MJ, Farver CF, Dweik RA, Kavuru MS, Erzurum SC, Hazen SL. Eosinophils generate brominating oxidants in allergen-induced asthma. J Clin Invest. 2000 May;105(10):1455-63. doi: 10.1172/JCI9702. PMID 10811853